CLINICAL TRIAL: NCT03575780
Title: A Phase 1 Open-label, Uncontrolled, Non-randomized, Maximal Use Pharmacokinetic Study to Evaluate the Systemic Exposure and Safety of KX2-391 Ointment 1% When Applied to 25 cm2 of the Face or Balding Scalp in Subjects With Actinic Keratosis
Brief Title: Single-Center Study Evaluating Systemic Exposure and Safety of KX2-391 Ointment 1% on the Face or Balding Scalp in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX01-AK-007
Record Dates: First submitted 2018-06-07; First posted 2018-07-03 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: This study will test KX2-391 Ointment 1%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KX2-391 Ointment (Experimental): KX2-391 ointment 1% will be administered once daily over 5 consecutive days
  Interventions: Drug: KX2-391 Ointment 1%

INTERVENTIONS:
Drug: KX2-391 Ointment 1% — The experimental drug, KX2-391 Ointment 1% will be used in subjects with Clinically typical Actinic Keratosis on the face or balding scalp.

SUMMARY:
This Phase I study is designed to evaluate the systemic exposure and safety of KX2-391 Ointment in adult subjects when applied to an area of skin containing at least 5 clinically typical, visible, and discrete Actinic Keratosis lesions on the face or balding scalp.

DETAILED DESCRIPTION:
This study will be a open-label, single center, pharmacokinetic, and safety study of KX2-391 Ointment administered topically to the face or balding scalp of subjects with actinic keratosis.

The study consists of Screening, Treatment, and Follow-up Periods. Eligible subjects will receive 5 consecutive days of topical treatment, to be applied at the same location. Activity (lesion counts) and safety evaluations will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years old.
2. Able to comprehend and are willing to sign an informed consent form (ICF).
3. At least 5 clinically typical, visible, and discrete AKs on 25 cm2 of the face or balding scalp.
4. Subjects who, in the judgment of the Investigator, are in good general health based on:

   1. Medical history
   2. Physical examination (PE) findings
   3. ECG, clinical chemistry, hematology, and urinalysis results.
5. In the case of a female of childbearing potential, TKL will initiate two forms of birth control at Screening and that at least one had to be in place for 30 days prior (oral/implant/injectable/transdermal contraceptives, intrauterine device (IUD), condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy, tubal ligation). Abstinence or vasectomies are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
6. Females of childbearing potential, must agree to continue to use two methods of birth control for 30 days following the last dose of study treatment;
7. In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) on Day 1 prior to randomization and are willing to submit to a UPT at the end of study (EOS);
8. In the case of sexually active males who have not had a vasectomy, and whose partner is reproductively capable, must agree to use barrier contraception from Screening through 90 days after their last dose of study treatment;
9. In the case of a female of non-childbearing potential, has had a hysterectomy or is postmenopausal (at least 2 years with no menses prior to enrollment);
10. All subjects must agree not to donate sperm or eggs or attempt conception from Screening through 90 days following their last dose of study treatment;
11. Willing to avoid direct sun or ultraviolet (UV) light exposure to the face or scalp.

Exclusion Criteria:

1. Clinically atypical and/or rapidly changing AK lesions on the treatment area, e.g., hypertrophic, hyperkeratotic, recalcitrant disease (had cryosurgery on two previous occasions) and/or cutaneous horn.
2. Location of the treatment area:

   1. Within 5 cm of an incompletely healed wound
   2. Within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
3. Been previously treated with KX2-391 ointment.
4. Has QTcF >450 ms for males and 470 ms for females or other relevant pathological changes in the ECG, in the opinion of the Investigation, at Screening.
5. Anticipated need for in-patient hospitalization or in-patient surgery during the study.
6. Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for AK within 2 cm of the treatment area, within 8 weeks prior to the Screening visit.
7. Use of the following therapies and/or medications within 2 weeks prior to the Screening visit:

   1. Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within 2 cm of the selected treatment area
   2. Acid-containing therapeutic products (e.g., salicylic acid or fruit acids, such as alpha- and beta-hydroxyl acids and glycolic acids), topical retinoids, or light chemical peels within 2 cm of the selected treatment area
   3. Topical salves (non-medicated/non-irritant lotion and cream are acceptable) or topical steroids within 2 cm of the selected treatment area; artificial tanners within 5 cm of the selected treatment area.
8. Use of the following therapies and/or medications within 4 weeks prior to the Screening visit:

   1. Treatment with immunomodulators (e.g., azathioprine), cytotoxic drugs (e.g., cyclophosphamide, vinblastine, chlorambucil, methotrexate) or interferons/interferon inducers
   2. Treatment with systemic medications that suppress the immune system (e.g., cyclosporine, prednisone, methotrexate, alefacept, infliximab)
   3. Therapy/treatment with UVA or UVB.
9. Use of systemic retinoids (e.g., isotretinoin, acitretin, bexarotene) within 6 months prior to the Screening visit.
10. A history of sensitivity and/or allergy to any of the ingredients in the study medication.
11. A skin disease (e.g., atopic dermatitis, psoriasis, eczema) or condition (e.g., scarring, open wounds) that, in the opinion of the Investigator, might interfere with the study conduct or evaluations, or which exposes the subject to unacceptable risk by study participation.
12. Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would exposure the subject to unacceptable risk by study participation.
13. Females who are pregnant or nursing.
14. Participated in an investigational drug trial during which an investigational study medication was administered within 30 days or 5 half-lives or the investigational product, whichever is longer, before dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Amount of KX2-391 Ointment in the blood stream | 6 Days
  The measurement of KX2-391 Ointment levels in the blood stream over time

SECONDARY OUTCOMES:
Local Skin Reactions | 29 Days
  To evaluate the safety of KX2-391 Ointment 1% by the proportion and severity of local skin reactions
Adverse Events | 29 Days
  To evaluate the safety of KX2-391 Ointment 1% by the proportion of adverse events
Abnormal Laboratory Assessments | 29 Days
  To evaluate the safety of KX2-391 Ointment 1% by the proportion of abnormal laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, FRCP, Study Chair — Athenex, Inc.
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided